CLINICAL TRIAL: NCT04298983
Title: Phase II Clinical Trial of Abemaciclib in Combination With Androgen Deprivation Therapy for Locally Advanced Prostate Cancer
Brief Title: Abemaciclib in Combination With Androgen Deprivation Therapy for Locally Advanced Prostate Cancer
Acronym: RAD 1805
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Abemaciclib efficacy
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Andrew McDonald, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300004706; I3Y-US-I001 (Other: Eli Lilly)
Record Dates: First submitted 2020-03-02; First posted 2020-03-06 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: abemaciclib; androgen deprivation therapy; radiation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — abemaciclib; Androgen Antagonists; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Abemaciclib + ADT+ RT (Experimental): Abemaciclib at 150 mg by mouth twice daily, androgen deprivation therapy (ADT), and radiation therapy in conjunction with ADT.
  Interventions: Drug: Abemaciclib 150 MG by mouth twice daily; Drug: Androgen deprivation therapy (ADT); Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Abemaciclib 150 MG by mouth twice daily — Abemaciclib will start with initiation of ADT, 3 months before RT, and pause 2 weeks prior to start of RT. Abemaciclib will resume with the first ADT administration post-radiation, which is about 1 month post radiation therapy. Abemaciclib will continue for a total of 24 months.
Drug: Androgen deprivation therapy (ADT) — ADT will be given every 3 months. ADT and Abemaciclib will pause 2 weeks prior to start of RT. ADT administration will resume with Abemaciclib post-radiation, which is about 1 month post radiation therapy. ADT will continue for a total of 24 months.
Radiation: Radiation Therapy — RT will start 3 months after initiation of ADT and Abemaciclib. RT will be given as standard of care- 180 cGy x 28 fractions to the whole pelvis and the prostate will receive 250 cGy x 28 fractions. After RT is completed, both ADT and Abemaciclib will resume and continue for 24 months.

SUMMARY:
This Phase II study is designed to study the clinical and radiologic response, as well as, safety and tolerability of abemaciclib in combination with androgen deprivation therapy (ADT) in patients with localized high-risk or locally advanced prostate cancer who are eligible for definitive radiation therapy (RT) and androgen deprivation therapy (ADT).

DETAILED DESCRIPTION:
A similar hormone-driven cancer akin to breast cancers is prostate cancer. These tumors are driven by androgen receptor signaling, and CDK4/6 has also been found to be a bona fide target pre-clinically for advanced prostate cancer cell models. Moreover, CDK4/6 inhibition can act as a radiation sensitizer through its effects on the DNA damage response and interactions with cell cycle pathway proteins. For example, it has been found that expression of DNA repair proteins can be regulated by E2F, a transcription factor necessary for the G1 to S phase transition. Also, cyclin D1 has been found to exert a direct role in DNA repair. Lastly, CDK4/6 inhibition has been found to modulate the DNA damage response. These data support the use of CDK4/6 inhibitors as a modulator of DNA damage to enhance sensitivity to radiation.

Given the role of CDK4/6 in tumor resistance to endocrine therapy, in activation of the DNA damage response, and in promoting radiation resistance, we hypothesize that the targeting of CDK4/6 with abemaciclib will enhance the cytotoxicity in combination with blockade of the androgen receptor pathway. Therefore, we propose a pilot phase II investigator initiated trial in patients with high-risk prostate cancer testing the tolerability and toxicity of abemaciclib in combination with ADT.

Patients will receive ADT for 2 years and will start 3 months before radiation therapy. Abemaciclib will start with initiation of ADT and pause 2 weeks prior to start of radiation therapy. Abemaciclib will resume with the first ADT administration post-radiation, which is about 1 month post radiation therapy. Abemaciclib and ADT will continue for a total ADT period of 24 months. Patients will receive study treatment until development of toxicity or disease progression on treatment or any reasons of withdrawal or a maximum of 24 months of therapy with ADT. Patients are seen every 4 weeks with laboratory evaluation. For toxicity or adverse events, patients will undergo labs, physical examination and grades of toxicities will be determined using NCI CTCAE version 4.03.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed (core biopsy proven) adenocarcinoma of prostate, localized high-risk or locally advanced.
* One of the below:

  * Gleason 7-8, any T-stage, and PSA > 20,
  * Gleason 8, ≥ T2, any PSA,
  * Gleason 9-10, any T-stage, any PSA
* Available biopsy of primary tumor or resected tumor specimen with adequate samples.
* Prior treatment with systemic anti-cancer agents is not allowed.
* ECOG PS=0 or 1.
* Must have at least 1 target lesion.
* Adequate hematologic and end-organ function:

  * ANC ≥ 1500/mm3
  * Platelet count ≥ 100,000/mm3
  * Hb ≥ 9g/dl
  * Creatinine ≤ ULN or Creatinine Clearance (CrCl) ≥ 60 ml/min
  * Total Bilirubin ≤ 1.5 x ULN (except subjects with Gilbert syndrome, who can have total Bilirubin > 2.0 x ULN and direct bilirubin within normal limits are permitted).
  * AST, ALT and alkaline phosphatase ≤ ULN
* Agreement to remain abstinent or use appropriate contraception.
* Willingness and ability to consent for self to participate in study.
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Prior treatment to CDK4-6 inhibitor.
* Prior treatment with systemic agents or radiation treatment for the primary cancer.
* Major surgical procedure or significant traumatic injury within 4 weeks prior to study treatment, and must have fully recovered from any such procedure.
* Personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
* Angina, myocardial infarction (MI), symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack (TIA), arterial embolism, pulmonary embolism, percutaneous transluminal coronary angioplasty (PTCA), or coronary artery bypass grafting (CABG) within 6 months prior to study treatment.
* Known active viral or non-viral hepatitis or cirrhosis.
* Any active infection requiring systemic treatment, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA).
* Known history of AIDS (acquired immunodeficiency syndrome)-defining illness.
* Patients must be surgically sterile or must agree to use effective contraception during the study treatment (including temporary breaks from treatment), and for at least 180 days after stopping last dose of Abemaciclib.
* Other severe and/or uncontrolled acute or chronic medical or psychiatric condition or laboratory abnormality that, in the judgment of the investigator, may increase the risk associated with study participation or may interfere with the interpretation of study results and would make the patient inappropriate for this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea.)
* Secondary malignancy requiring active treatment. Past history of malignancy other than prostate cancer treated with curative intent and not requiring additional treatment may be eligible after discussion with PI.
* Patients with active autoimmune disease and history of inflammatory bowel disease. Brachytherapy boost will not be permitted.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McDonald, MD, Principal Investigator — University of Alabama at Birmingham (UAB)
Locations (1):
- University of Alabama at Birmingham (UAB), Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abemaciclib + ADT+ RT
Started | 9
Completed | 2
Not Completed | 7
Not completed — Adverse Event | 4
Not completed — Lack of Efficacy | 3

BASELINE CHARACTERISTICS:
Arm/Group | Abemaciclib + ADT+ RT
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Clinical Response Rates
Description: Clinical response rates will be assessed by percentage of patients who achieve the PSA nadir levels of < 0.5ng/ml on treatment
Time Frame: Baseline to 24 months
Population: A total of 9 patients were enrolled in the study. Two patients completed the entire protocol specified therapy. Both of these patients achieved clinical response. 4 patients were taken off study drug due to SAEs. The trial was terminated (along with the 3 remaining patients discontinuing drug) early due to negative results of a later phase clinical trial in men with metastatic prostate cancer.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib + ADT+ RT
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Number of Patients With PSA Declines Prior to Radiotherapy
Description: Number of patients with PSA declines prior to radiotherapy- calculated from nadir level prior to initiation of radiation therapy
Time Frame: Up to 3 months of treatment
Population: A total of 9 patients were enrolled in the study. Two patients completed the entire protocol specified therapy. Both patients had PSA declines prior to radiotherpay. 4 patients were taken off study drug due to SAEs. The trial was terminated (along with the 3 remaining patients discontinuing drug) early due to negative results of a later phase clinical trial in men with metastatic prostate cancer.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib + ADT+ RT
Number analyzed (Participants) | 2
Participants | 2

3. Secondary Outcome: Number of Patients to Experience PSA Failure
Description: Number of patients to experience PSA failure will be analyzed using the Kaplan-Meier method
Time Frame: Baseline up to 24 months
Population: A total of 9 patients were enrolled in the study. Two patients completed the entire protocol specified therapy. The two patients were analyzed and neither experienced PSA failure. 4 patients were taken off study drug due to SAEs. The trial was terminated (along with the 3 remaining patients discontinuing drug) early due to negative results of a later phase clinical trial in men with metastatic prostate cancer.
Measure: Count of Participants; unit: Participants
Arm/Group | Abemaciclib + ADT+ RT
Number analyzed (Participants) | 2
Participants | 0

ADVERSE EVENTS:
Time Frame: Each participant was assessed up to 24 months.
Arm/Group | Abemaciclib + ADT+ RT
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 4/9
Other Adverse Events (participants affected / at risk) | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abemaciclib + ADT+ RT (N=9)
Lipase Increased (Investigations) | 4

LIMITATIONS AND CAVEATS:
A total of 9 patients were enrolled in the study. Two patients completed the entire protocol specified therapy. 4 patients were taken off study drug due to SAEs. The trial was terminated (along with the 3 remaining patients discontinuing drug) early due to negative results of a later phase clinical trial in men with metastatic prostate cancer. No longer proceeding with study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/83/NCT04298983/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/83/NCT04298983/ICF_001.pdf